CLINICAL TRIAL: NCT02106832
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Study Comparing Ciprofloxacin DPI 32.5 mg BID (Twice a Day) Intermittently Administered for 28 Days on / 28 Days Off or 14 Days on / 14 Days Off Versus Placebo to Evaluate the Time to First Pulmonary Exacerbation and Frequency of Exacerbations in Subjects With Non-Cystic Fibrosis Bronchiectasis.
Brief Title: Ciprofloxacin Dry Powder for Inhalation (DPI) in Non-cystic Fibrosis Bronchiectasis (Non-CF BE)
Acronym: RESPIRE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15626; 2013-004659-19 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Bronchiectasis
Keywords: Ciprofloxacin; Dry Powder for Inhalation; Exacerbation; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Ciprofloxacin; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ciprofloxacin DPI 28 Days on/off (Cipro 28) (Experimental): Subjects received ciprofloxacin (BAYQ3939) 32.5 milligram (mg) corresponding to 50 mg dry powder for inhalation (DPI) administered twice daily (BID) (every 12 hours); a treatment cycle consisted of a 28-day on-treatment phase followed by a 28-day off-treatment phase (48 weeks treatment phase = 6 active cycles).
  Interventions: Drug: Ciprofloxacin (BAYQ3939) dry powder for inhalation
- Ciprofloxacin DPI 14 Days on/off (Cipro 14) (Experimental): Subjects received ciprofloxacin 32.5 mg corresponding to 50 mg DPI administered BID (every 12 hours); a treatment cycle consisted of a 14-day on-treatment phase followed by a 14-day off-treatment phase (48 weeks treatment phase = 12 active cycles).
  Interventions: Drug: Ciprofloxacin (BAYQ3939) dry powder for inhalation
- Placebo 28 Days on/off (Placebo 28) (Placebo Comparator): Subjects received placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of a 28-day on-treatment phase followed by a 28-day off-treatment phase (48 weeks treatment phase = 6 cycles).
  Interventions: Drug: Placebo
- Placebo 14 Days on/off (Placebo 14) (Placebo Comparator): Subjects received placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of a 14-day on-treatment phase followed by a 14-day off-treatment phase (48 weeks treatment phase = 12 cycles).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin (BAYQ3939) dry powder for inhalation — Ciprofloxacin dry powder for inhalation (DPI) 32.5 mg inhaled twice daily in cycles of 28 days on-treatment and 28 days off-treatment.
  Arms: Ciprofloxacin DPI 28 Days on/off (Cipro 28)
Drug: Ciprofloxacin (BAYQ3939) dry powder for inhalation — Ciprofloxacin DPI 32.5 mg inhaled twice daily in cycles of 14 days on-treatment and 14 days off-treatment.
  Arms: Ciprofloxacin DPI 14 Days on/off (Cipro 14)
Drug: Placebo — Matching placebo inhaled twice daily intermittently for 28 days on / 28 days off
  Arms: Placebo 28 Days on/off (Placebo 28)
Drug: Placebo — Matching placebo inhaled twice daily intermittently for 14 days on / 14 days off
  Arms: Placebo 14 Days on/off (Placebo 14)

SUMMARY:
The purpose of this study is to evaluate if the time to first pulmonary exacerbation of bronchiectasis or its frequency can be prolonged by inhalation of ciprofloxacin for 28 days every other 28 days or for 14 days every other 14 days over 48 weeks.

DETAILED DESCRIPTION:
Number of participants with Adverse events will be covered in Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a proven and documented diagnosis of non CF idiopathic or post infectious bronchiectasis
* Stable pulmonary status and stable regimen of standard treatment at least for the past 4 weeks

Exclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) <30% or >90% predicted
* Active allergic bronchopulmonary aspergillosis
* Active and actively treated non tuberculosis mycobacterial (NTM) infection or tuberculosis
* Primary diagnosis of Chronic obstructive pulmonary disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (169):
- United States (22):
  - Peoria, Arizona
  - Fountain Valley, California
  - La Jolla, California
  - Long Beach, California
  - Newport Beach, California
  - San Diego, California
  - Kissimmee, Florida
  - Miami, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Skokie, Illinois
  - Olathe, Kansas
  - Rochester, Minnesota
  - Brooklyn, New York
  - Mineola, New York
  - Asheville, North Carolina
  - Portland, Oregon
  - Doylestown, Pennsylvania
  - Greenville, South Carolina
  - Edinburg, Texas
  - Tyler, Texas
- Argentina (5):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Capital Federal, Ciudad Auton. de Buenos Aires
  - Godoy Cruz, Mendoza Province
  - Córdoba
  - Vicente López
- Australia (6):
  - Kogarah, New South Wales
  - New Lambton Heights, New South Wales
  - Adelaide, South Australia
  - Parkville, Victoria
  - Murdoch, Western Australia
  - Perth, Western Australia
- Austria (2):
  - Graz
  - Salzburg
- Brazil (6):
  - Belo Horizonte, Minas Gerais
  - Recife, Pernambuco
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Porto Alegre
  - São Paulo
- Bulgaria (9):
  - Gabrovo
  - Kozloduy
  - Lovech
  - Razgrad
  - Rousse
  - Sevlievo
  - Sliven
  - Sofia
  - Stara Zagora
- China (12):
  - Fuzhou, Fujian
  - Guangzhou, Guangdong
  - Hohehot, Inner Mongolia
  - Suzhou, Jiangsu
  - Wuxi, Jiangsu
  - Nanchang, Jiangxi
  - Shenyang, Liaoning
  - Yinchuan, Ningxia
  - Chengdu, Sichuan
  - Beijing
  - Chongqing
  - Shanghai
- Czechia (2):
  - Brno
  - Prague
- Germany (10):
  - Treuenbrietzen, Brandenburg
  - Frankfurt am Main, Hesse
  - Neu-Isenburg, Hesse
  - Hanover, Lower Saxony
  - Gelsenkirchen, North Rhine-Westphalia
  - Leipzig, Saxony
  - Bad Berka, Thuringia
  - Jena, Thuringia
  - Berlin
  - Hamburg
- Hong Kong (4):
  - Hong Kong
  - Kowloon
  - New Territories
  - Shatin
- Latvia (5):
  - Daugavpils
  - Jūrmala
  - Krāslava
  - Riga
  - Talsi
- Lithuania (2):
  - Klaipėda
  - Vilnius
- Netherlands (7):
  - Alkmaar
  - Assen
  - Groningen
  - Helmond
  - Maastricht
  - Sittard-Geleen
  - Veldhoven
- Philippines (3):
  - City of San Fernando
  - Manila
  - Quezon City
- Poland (12):
  - Bielsko-Biala
  - Częstochowa
  - Gorzów Wielkopolski
  - Grudziądz
  - Katowice
  - Kielce
  - Krakow
  - Ksawerów
  - Mrozy
  - Ostrowiec Świętokrzyski
  - Rzeszów
  - Warsaw
- Portugal (4):
  - Angra do Heroísmo, Azores
  - Vila Nova de Gaia, Porto District
  - Faro
  - Lisbon
- Romania (8):
  - Bragadiru
  - Brasov
  - Bucharest
  - Codlea
  - Constanța
  - Iași
  - Ploieşti
  - Timișoara
- Russia (10):
  - Arkhangelsk
  - Chelyabinsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Saint Petersburg
  - Tomsk
  - Ufa
  - Voronezh
  - Yaroslavl
- Serbia (7):
  - Belgrade
  - Čačak
  - Kamenitz
  - Knez-Selo
  - Kragujevac
  - Sombor
  - Valjevo
- Slovakia (2):
  - Bratislava
  - Prešov
- South Africa (3):
  - Johannesburg, Gauteng
  - eManzimtoti, KwaZulu-Natal
  - Cape Town, Western Cape
- South Korea (7):
  - Daejeon, Daejeon Gwang''yeogsi
  - Bucheon-si, Gyeonggido
  - Incheon Gwangyeogsi,, Incheon Gwang''yeogsi
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Incheon
  - Seoul
- Taiwan (5):
  - Chiayi City
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei
- Thailand (6):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - NakhonRatchasima
  - Phitsanulok
  - Udon Thani
- Turkey (Türkiye) (10):
  - Ankara
  - Balcalı
  - Izmir
  - Kampus
  - Konya
  - Maltepe
  - Mersin
  - Pendik
  - Samsun
  - Şehitkamil

REFERENCES:
- [Derived] Aksamit T, De Soyza A, Bandel TJ, Criollo M, Elborn JS, Operschall E, Polverino E, Roth K, Winthrop KL, Wilson R. RESPIRE 2: a phase III placebo-controlled randomised trial of ciprofloxacin dry powder for inhalation in non-cystic fibrosis bronchiectasis. Eur Respir J. 2018 Jan 25;51(1):1702053. doi: 10.1183/13993003.02053-2017. Print 2018 Jan. PMID 29371384
- [Derived] Aksamit T, Bandel TJ, Criollo M, De Soyza A, Elborn JS, Operschall E, Polverino E, Roth K, Winthrop KL, Wilson R. The RESPIRE trials: Two phase III, randomized, multicentre, placebo-controlled trials of Ciprofloxacin Dry Powder for Inhalation (Ciprofloxacin DPI) in non-cystic fibrosis bronchiectasis. Contemp Clin Trials. 2017 Jul;58:78-85. doi: 10.1016/j.cct.2017.05.007. Epub 2017 May 8. PMID 28495619
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 164 study centers in 25 countries between 30 April 2014 (first subject first visit) and 19 October 2016 (last subject last visit).
Pre-assignment Details: A total of 1123 subjects were screened and 521 subjects were randomized. The randomized subjects were allocated to treatment groups, and 2 subjects in the Cipro 14 group did not receive study medication.
Period: Overall Study
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Started | 171 | 176 | 86 | 88
Participants Received Treatment | 171 | 174 | 86 | 88
Completed | 148 | 151 | 70 | 73
Not Completed | 23 | 25 | 16 | 15
Not completed — Adverse Event | 1 | 2 | 3 | 0
Not completed — Death | 4 | 4 | 1 | 4
Not completed — Deterioration of general conditions | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 17 | 17 | 10 | 7
Not completed — Technical problems | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14) | Total
Number analyzed (Participants) | 171 | 176 | 86 | 88 | 521
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (14.2) | 60.4 (13.7) | 60.6 (13.7) | 60.4 (15.0) | 60.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 96 | 52 | 62 | 302
  Male | 79 | 80 | 34 | 26 | 219
Saint George's Respiratory Questionnaire (SGRQ) Symptoms Component Score [Mean (Standard Deviation); unit: Score on a scale] — The SGRQ was a validated, disease-specific instrument that measures health-related quality of life (HRQoL) in adults with chronic obstructive pulmonary disease (COPD) and asthma and was later validated for use in bronchiectasis. The SGRQ covers 3 dimensions: symptoms, activity and impact on daily life. To determine the outcome, a score ranging from 1 to 100 was calculated for each individual domain and for the total score, and smaller scores indicate better health status. For this baseline measure, the symptoms component score was reported.
  Score on a scale | 60.75 (20.61) | 61.26 (19.54) | 58.56 (19.17) | 63.47 (19.48) | 61.00 (19.82)
Quality of Life Questionnaire for Bronchiectasis (QoL-B) Respiratory Symptoms Domain Score [Mean (Standard Deviation); unit: Score on a scale] — The QoL-B was a disease-specific questionnaire developed for non-Cystic fibrosis Bronchiectasis. It covers 8 dimensions: physical functioning, role functioning, emotional functioning, social functioning, vitality, treatment burden, health perceptions, and respiratory symptoms. Each dimension was scored separately on a scale of 0 to 100, and higher scores represent better outcomes. For this baseline measure, the respiratory symptoms domain score was reported.
  Score on a scale | 50.14 (19.07) | 52.17 (18.49) | 53.95 (16.00) | 48.67 (17.72) | 51.22 (18.16)
Forced Expiratory Volume in One Second (FEV1) [Mean (Standard Deviation); unit: Liter] — FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters at body temperature and ambient pressure saturated with water vapor (BTPS).
  Liter | 1.569 (0.602) | 1.519 (0.617) | 1.560 (0.692) | 1.477 (0.558) | 1.535 (0.615)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Exacerbation Event Within 48 Weeks - Cipro 28 vs. Pooled Placebo
Description: Time to first exacerbation was defined as the time from randomization until the visit at which the first qualifying exacerbation is recorded by the investigator. Exacerbation events are defined as exacerbations with systemic antibiotic use and presence of fever or malaise / fatigue and worsening of at least three signs/symptoms.
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Median (99.9% Confidence Interval); unit: Days
Groups:
- Pooled Placebo: Subjects received matching placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of either a 28-day days on-treatment phase followed by 28-day off-treatment phase or 14-day on-treatment phase followed by 14-day off treatment phase (48 weeks treatment phase = 6 cycles and 12 cycles, respectively).
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Pooled Placebo
Number analyzed (Participants) | 171 | 174
Days | NA [NA to NA] — Value cannot be estimated due to censored data. | NA [211 to NA] — Value cannot be estimated due to censored data.
Statistical Analysis 1: Comparison: Ciprofloxacin DPI 28 Days on/Off (Cipro 28) vs Pooled Placebo; The hazard ratio for time to first exacerbation event within 48 weeks and 99.9% Confidence Interval (CI) was calculated by using Cox proportional hazards model by comparison of Cipro 28/Pooled Placebo reporting groups. P-value was analysed using Wald-type test; Test type: Superiority or Other; p = 0.0511, Wald-type test; Hazard Ratio (HR) = 0.7062, 99.9% CI 2-sided [0.3928 to 1.2698]

2. Secondary Outcome: Number of Participants With Exacerbation Events With Worsening of at Least Three Signs/Symptoms Over 48 Weeks
Description: For this outcome measure, exacerbation events were defined as exacerbations with systemic antibiotic use and presence of fever or malaise / fatigue and worsening of at least three signs/symptoms over 48 weeks.
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 171 | 176 | 174
Participants
  Number of exacerbations: 0 | 115 | 108 | 101
  Number of exacerbations: 1 | 46 | 40 | 41
  Number of exacerbations: 2 | 8 | 23 | 19
  Number of exacerbations: 3 | 2 | 4 | 10
  Number of exacerbations: 4 | 0 | 1 | 2
  Number of exacerbations: 5 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Exacerbation Events With Worsening of at Least One Sign/Symptom Over 48 Weeks
Description: For this outcome measure, exacerbation events were defined as exacerbations with systemic antibiotic use and worsening of at least one sign/symptom over 48 weeks.
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 171 | 176 | 174
Participants
  Number of exacerbations: 0 | 102 | 96 | 90
  Number of exacerbations: 1 | 51 | 46 | 45
  Number of exacerbations: 2 | 14 | 26 | 22
  Number of exacerbations: 3 | 3 | 4 | 11
  Number of exacerbations: 4 | 1 | 3 | 4
  Number of exacerbations: 5 | 0 | 1 | 2

4. Secondary Outcome: Percentage of Participants With Pathogen Eradication at End of Treatment (Week 44/46)
Description: Pathogen eradication was defined as a negative culture result for all pre-specified pathogens at end of treatment (week 44 or 46 depending on treatment regimen) that were present in the participant at baseline. There was no imputation for participants who discontinued the study prematurely.
Time Frame: End of treatment (Week 44/46)
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 171 | 176 | 174
Percentage of participants
  No | 35.1 | 35.8 | 40.2
  Yes | 31.6 | 35.8 | 31.6

5. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcome Saint George's Respiratory Questionnaire (SGRQ) Symptoms Component Score at End of Treatment (Week 44/46)
Description: The SGRQ was a validated, disease-specific instrument that measures health-related quality of life (HRQoL) in adults with chronic obstructive pulmonary disease (COPD) and asthma and was later validated for use in bronchiectasis. The SGRQ covers 3 dimensions: symptoms, activity and impact on daily life. To determine the outcome, a score ranging from 1 to 100 was calculated for each individual domain and for the total score, and smaller scores indicate better health status. For this outcome measure, the symptoms component score was reported.
Time Frame: Baseline and end of treatment (Week 44/46)
Population: FAS with participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Number analyzed (Participants) | 142 | 142 | 67 | 72
Score on a scale | -8.92 (21.06) | -9.02 (20.10) | -2.91 (24.48) | -11.50 (18.54)

6. Secondary Outcome: Percentage of Participants With Occurrence of New Pathogens Present at End of Treatment (Week 44/46)
Description: New pathogens were any of the pre-specified organisms not cultured before start of study medication. There was no imputation for participants who discontinued the study prematurely.
Time Frame: End of treatment (Week 44/46)
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 171 | 176 | 174
Percentage of participants
  No | 62.6 | 67.6 | 61.5
  Yes | 4.1 | 4.0 | 10.3

7. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcome Quality of Life Questionnaire for Bronchiectasis (QoL-B) Respiratory Symptoms Domain Score at End of Treatment (Week 44/46)
Description: The QoL-B was a disease-specific questionnaire developed for non-Cystic fibrosis Bronchiectasis. It covers 8 dimensions: physical functioning, role functioning, emotional functioning, social functioning, vitality, treatment burden, health perceptions, and respiratory symptoms. Each dimension was scored separately on a scale of 0 to 100, and higher scores represent better outcomes. For this outcome measure, the respiratory symptoms domain score was reported.
Time Frame: Baseline and end of treatment (Week 44/46)
Population: FAS with participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Number analyzed (Participants) | 85 | 94 | 43 | 49
Score on a scale | 11.57 (17.49) | 10.90 (18.07) | 7.08 (17.00) | 10.70 (15.58)

8. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at End of Treatment (Week 44/46)
Description: FEV1 was defined as the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters at body temperature and ambient pressure saturated with water vapor (BTPS).
Time Frame: Baseline and end of treatment (Week 44/46)
Population: FAS with participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Number analyzed (Participants) | 138 | 140 | 62 | 71
Liter | 0.038 (0.336) | -0.037 (0.287) | -0.038 (0.272) | 0.037 (0.299)

9. Primary Outcome: Time to First Exacerbation Event Within 48 Weeks - Cipro 14 vs. Pooled Placebo
Description: as for outcome 1
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Median (95.1% Confidence Interval); unit: Days
Arm/Group | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 176 | 174
Days | NA [NA to NA] — Value cannot be estimated due to censored data. | NA [278 to NA] — Value cannot be estimated due to censored data.
Statistical Analysis 1: Comparison: Ciprofloxacin DPI 14 Days on/Off (Cipro 14) vs Pooled Placebo; The hazard ratio for time to first exacerbation event within 48 weeks and 95.1% Confidence Interval (CI) was calculated by using Cox proportional hazards model by comparison of Cipro 28/Pooled Placebo reporting groups. P-value was analysed using Wald-type test; Test type: Superiority or Other; p = 0.3965, Wald-type test; Hazard Ratio (HR) = 0.8662, 95.1% CI 2-sided [0.6206 to 1.2090]

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after the last study drug administration.
Groups:
- Ciprofloxacin DPI 28 Days on/Off (Cipro 28): Subjects received ciprofloxacin (BAYQ3939) 32.5 mg corresponding to 50 mg DPI administered BID (every 12 hours); a treatment cycle consisted of a 28-day on-treatment phase followed by a 28-day off-treatment phase (48 weeks treatment phase = 6 active cycles).
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Serious Adverse Events (participants affected / at risk) | 28/171 | 45/174 | 41/174
Other Adverse Events (participants affected / at risk) | 51/171 | 60/174 | 55/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) (N=171) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) (N=174) | Pooled Placebo (N=174)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4) | 2 (2) | 2 (2)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 3 (3) | 2 (4)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 24 (27) | 21 (31)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) (N=171) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) (N=174) | Pooled Placebo (N=174)
Nasopharyngitis (Infections and infestations) | 10 (11) | 16 (19) | 14 (18)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 8 (10) | 5 (6)
Dysgeusia (Nervous system disorders) | 9 (13) | 8 (16) | 2 (2)
Headache (Nervous system disorders) | 10 (15) | 10 (11) | 5 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 7 (7) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (11) | 3 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 (19) | 15 (22) | 20 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer acknowledges and accepts the interest in the non-commercial scientific publication of Results. In a multi-center study the Principal Investigators will not make any publication of the results before the first multi-center publication. Proposed publication/presentation shall be provided to Bayer at least 60 days prior to the intended submission or presentation of the publication in order to allow Bayer to review it. Any difference of opinion shall be discussed.